CLINICAL TRIAL: NCT04388670
Title: Epidemiological and Clinical Characteristics of Patients With COVID-19 Admitted in Italian Intensive Care Units: a Multicentric Retrospective-prospective Cohort Study.
Brief Title: Epidemiological and Clinical Characteristics of Critically Ill Patients With COVID-19
Acronym: 2019nCoV_ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Associate Professor, Policlinico Hospital
Other Study IDs: PoliclinicoH
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Critical Illness
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective of this observational multicentric retrospective-prospective study is to describe the number and the characteristics of patients with Reverse Transcription Polymerase Chain Reaction (RT-PCR) for SARS-CoV2 positivity admitted to Intensive Care Units during the first 6 months of epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Adulthood
* Informed consent obtained

Exclusion Criteria:

* No informed consent obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with COVID-19 admitted in Intensive Care Units.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-02-22 (Actual); Primary Completion 2020-08-22 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall number and characteristics of patients with COVID-19 in ICU | 22nd February - 22nd August 2020
  Number and characteristics of patients with COVID-19 admitted in Intensive Care Units every week.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Grasselli, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Derived] Protti A, Madotto F, Florio G, Bove T, Carlesso E, Casella G, Dalla Corte F, Foti G, Giudici R, Langer T, Montalto C, Rezoagli E, Santini A, Terragni P, Zanella A, Grasselli G, Cecconi M. A tidal volume of 7 mL/kg PBW or higher may be safe for COVID-19 patients. J Crit Care. 2025 Feb;85:154921. doi: 10.1016/j.jcrc.2024.154921. Epub 2024 Sep 25. PMID 39326356
- [Derived] Scaravilli V, Guzzardella A, Madotto F, Beltrama V, Muscatello A, Bellani G, Monti G, Greco M, Pesenti A, Bandera A, Grasselli G. Impact of dexamethasone on the incidence of ventilator-associated pneumonia in mechanically ventilated COVID-19 patients: a propensity-matched cohort study. Crit Care. 2022 Jun 13;26(1):176. doi: 10.1186/s13054-022-04049-2. PMID 35698155
- [Derived] Zanella A, Florio G, Antonelli M, Bellani G, Berselli A, Bove T, Cabrini L, Carlesso E, Castelli GP, Cecconi M, Citerio G, Coloretti I, Corti D, Dalla Corte F, De Robertis E, Foti G, Fumagalli R, Girardis M, Giudici R, Guiotto L, Langer T, Mirabella L, Pasero D, Protti A, Ranieri MV, Rona R, Scudeller L, Severgnini P, Spadaro S, Stocchetti N, Vigano M, Pesenti A, Grasselli G; COVID-19 Italian ICU Network. Time course of risk factors associated with mortality of 1260 critically ill patients with COVID-19 admitted to 24 Italian intensive care units. Intensive Care Med. 2021 Sep;47(9):995-1008. doi: 10.1007/s00134-021-06495-y. Epub 2021 Aug 9. PMID 34373952
- [Derived] Grasselli G, Scaravilli V, Mangioni D, Scudeller L, Alagna L, Bartoletti M, Bellani G, Biagioni E, Bonfanti P, Bottino N, Coloretti I, Cutuli SL, De Pascale G, Ferlicca D, Fior G, Forastieri A, Franzetti M, Greco M, Guzzardella A, Linguadoca S, Meschiari M, Messina A, Monti G, Morelli P, Muscatello A, Redaelli S, Stefanini F, Tonetti T, Antonelli M, Cecconi M, Foti G, Fumagalli R, Girardis M, Ranieri M, Viale P, Raviglione M, Pesenti A, Gori A, Bandera A. Hospital-Acquired Infections in Critically Ill Patients With COVID-19. Chest. 2021 Aug;160(2):454-465. doi: 10.1016/j.chest.2021.04.002. Epub 2021 Apr 20. PMID 33857475
- [Derived] Langer T, Brioni M, Guzzardella A, Carlesso E, Cabrini L, Castelli G, Dalla Corte F, De Robertis E, Favarato M, Forastieri A, Forlini C, Girardis M, Grieco DL, Mirabella L, Noseda V, Previtali P, Protti A, Rona R, Tardini F, Tonetti T, Zannoni F, Antonelli M, Foti G, Ranieri M, Pesenti A, Fumagalli R, Grasselli G; PRONA-COVID Group. Prone position in intubated, mechanically ventilated patients with COVID-19: a multi-centric study of more than 1000 patients. Crit Care. 2021 Apr 6;25(1):128. doi: 10.1186/s13054-021-03552-2. PMID 33823862